CLINICAL TRIAL: NCT03577054
Title: Development of a Mobile Application Through User Centered Design to Improve Helping Babies Breath Skills Retention
Brief Title: Development of a Mobile Application for HBB Prompt Study
Acronym: HBB-Prompt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MUST 16/09-17
Record Dates: First submitted 2018-05-15; First posted 2018-07-05 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Birth Asphyxia; Neonatal Death
Keywords: Helping Babies Breathe; newborn resuscitation; skills retention; mobile health; user-centred design
MeSH Terms: conditions — Asphyxia Neonatorum; Perinatal Death

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor at analysis stage will be masked to allocation of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBB Prompt (Experimental): The investigators will train frontline health providers in Helping Babies Breathe (HBB) 2.0 and Essential Care for Every Baby (ECEB). Providers will undergo ECEB training in addition to HBB as these training programs are recommended by the Uganda Ministry of Health to be offered together.
  Providers at this hospital will have access to the most updated version of HBB Prompt (beta) after HBB training.
  Participants in will be asked to achieve a minimum practice target of once per day (low-dose high frequency training). The recommended frequency to use the app will be once per shift.
  Interventions: Behavioral: HBB Prompt; Behavioral: Low-Dose High Frequency training
- Control (Placebo Comparator): The investigators will train frontline health providers in Helping Babies Breathe (HBB) 2.0 and Essential Care for Every Baby (ECEB). Providers will undergo ECEB training in addition to HBB as these training programs are recommended by the Uganda Ministry of Health to be offered together.
  The control group will not have exposure to the HBB Prompt app post training. Participants in will be asked to achieve a minimum practice target of once per day (low-dose high frequency training).
  Interventions: Behavioral: Low-Dose High Frequency training

INTERVENTIONS:
Behavioral: HBB Prompt — Mobile app developed through user-centred design in phase 1 of this study
  Other Names: mobile app
  Arms: HBB Prompt
Behavioral: Low-Dose High Frequency training — Participants will be encouraged to practice their HBB skills daily
  Other Names: LDHF

SUMMARY:
This study applies an iterative user-centred design approach involving frontline birth attendants to create a mobile application ("HBB Prompt") to improve skills retention after initial newborn stabilization training through the Helping Babies Breathe (HBB) program. HBB Prompt will then be piloted at one site after HBB training and skills retention will be compared with a control site without HBB Prompt after HBB training.

DETAILED DESCRIPTION:
Helping Babies Breathe (HBB) is a newborn stabilization course that has been shown to reduce neonatal mortality by up to 47%. Such mortality impact is however not sustained due to rapid skills deterioration.

The investigators propose to improve sustainability of HBB's impact by increasing skills retention with an innovative mobile application called HBB Prompt. HBB Prompt will be an interactive tool that guides frontline providers through the steps needed to save newborn babies at birth. HBB Prompt will facilitate individual and group training in health facilities using the Low Dose High Frequency model (LDHF) for resuscitation skills retention.

The investigators will robustly develop HBB Prompt by integrating human factors and user-centered design approaches. The investigators will engage end-users and HBB Master Trainers to iteratively collect feedback to develop HBB Prompt for both individual and small group resuscitation practice. The iterative approach will mitigate the common scenario of mobile health (mHealth) solutions unable to achieve sustained success at scale due to lack of comprehensive input from frontline users.

The investigators will pilot the app at a single centre and compare it to a control site for HBB skills retention at different time points after initial HBB training.

ELIGIBILITY:
Inclusion Criteria:

* Frontline birth attendants involved in the delivery or care of babies in the maternity ward, theater or pediatric wards with a possibility of involvement in newborn resuscitation.

Exclusion Criteria:

* Health workers providing care in other wards other than maternity and pediatrics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Helping Babies Breathe Objective Structured Clinical Exam (OSCE) B score | 12 months from initial HBB training
  standardized comprehensive evaluation of HBB skills, 17 out of 23 constitutes a pass score with 23 being the highest score. The OSCE B is a standard Helping Babies Breathe assessment tool that comprises the steps required in successfully assisting a neonate in its transition after birth

SECONDARY OUTCOMES:
OSCE B score | immediately before initial HBB training
  standardized comprehensive evaluation of HBB skills, 17 out of 23 constitutes a pass score
OSCE B score | immediately after initial HBB training
  standardized comprehensive evaluation of HBB skills, 17 out of 23 constitutes a pass score
OSCE B score | 3 months from initial HBB training
  standardized comprehensive evaluation of HBB skills, 17 out of 23 constitutes a pass score
OSCE B score | 6 months from initial HBB training
  standardized comprehensive evaluation of HBB skills, 17 out of 23 constitutes a pass score
HBB 2.0 Knowledge Check | at unannounced visits within 12 months of training
  18 questions pertaining to newborn resuscitation
Bag and mask ventilation skills check | at unannounced visits within 12 months of training
  evaluation of bagging skills to assist breathing - score out of 14
Bag and mask ventilation quality measures with AIR Device | at unannounced visits within 12 months of training
  Augmented Infant Resuscitator (AIR) to objectively measure quality of newborn resuscitation during every ventilation epoch. AIR records time stamped data on ventilation quality, such as presence of air leak or obstruction and ventilation rate (www.air-device.com)
OSCE A | at unannounced visits within 12 months of training
  standardized evaluation of resuscitation skills (slightly different scenario than for OSCE B), 9 out of 12 constitutes a pass score
App analytics - pattern of usage | during 12 months after initial training in intervention arm only
  automated reports from the app regarding usage of different components of the app
App analytics - frequency of usage | during 12 months after initial training in intervention arm only
  frequency of access to different parts of the app, duration of app usage
App analytics - trends of performance | during 12 months after initial training in intervention arm only
  time trends of knowledge checks and simulation evaluations as noted in the app
Frequency of practice | during 12 months after initial training
  for both intervention and control arms, log-books will be reviewed for frequency of practice and in the intervention arm, this will be compared to what is reported through the app
Exit focus group feedback on barriers and facilitators to HBB training and skills maintenance | at end of study (12 months from the start)
  both intervention and control group participants will be interviewed to provide feedback on facilitators and barriers to HBB skills maintenance, and in the intervention arm, whether HBB Prompt helped or hindered their skills maintenance

OTHER OUTCOMES:
Delivery Volume | during 12 month study period
  number of births will be recorded from the birth register of each site
Infants requiring bagging | during 12 month study period
  number of babies requiring bagging will be recorded from the birth register of each site
Fresh stillbirths | during 12 month study period
  number of fresh stillbirths will be recorded from the birth register of each site
In hospital neonatal mortality | during 12 month study period
  number of neonatal deaths prior to discharge will be recorded from the birth register of each site

CONTACTS AND LOCATIONS:
Overall Officials: Santorino Data, MBChB, MMed, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Msemo G, Massawe A, Mmbando D, Rusibamayila N, Manji K, Kidanto HL, Mwizamuholya D, Ringia P, Ersdal HL, Perlman J. Newborn mortality and fresh stillbirth rates in Tanzania after helping babies breathe training. Pediatrics. 2013 Feb;131(2):e353-60. doi: 10.1542/peds.2012-1795. Epub 2013 Jan 21. PMID 23339223
- [Background] Kc A, Wrammert J, Clark RB, Ewald U, Vitrakoti R, Chaudhary P, Pun A, Raaijmakers H, Malqvist M. Reducing Perinatal Mortality in Nepal Using Helping Babies Breathe. Pediatrics. 2016 Jun;137(6):e20150117. doi: 10.1542/peds.2015-0117. PMID 27225317
- [Background] Goudar SS, Somannavar MS, Clark R, Lockyer JM, Revankar AP, Fidler HM, Sloan NL, Niermeyer S, Keenan WJ, Singhal N. Stillbirth and newborn mortality in India after helping babies breathe training. Pediatrics. 2013 Feb;131(2):e344-52. doi: 10.1542/peds.2012-2112. Epub 2013 Jan 21. PMID 23339215
- [Background] Bang A, Patel A, Bellad R, Gisore P, Goudar SS, Esamai F, Liechty EA, Meleth S, Goco N, Niermeyer S, Keenan W, Kamath-Rayne BD, Little GA, Clarke SB, Flanagan VA, Bucher S, Jain M, Mujawar N, Jain V, Rukunga J, Mahantshetti N, Dhaded S, Bhandankar M, McClure EM, Carlo WA, Wright LL, Hibberd PL. Helping Babies Breathe (HBB) training: What happens to knowledge and skills over time? BMC Pregnancy Childbirth. 2016 Nov 22;16(1):364. doi: 10.1186/s12884-016-1141-3. PMID 27875999
- [Background] Reisman J, Arlington L, Jensen L, Louis H, Suarez-Rebling D, Nelson BD. Newborn Resuscitation Training in Resource-Limited Settings: A Systematic Literature Review. Pediatrics. 2016 Aug;138(2):e20154490. doi: 10.1542/peds.2015-4490. Epub 2016 Jul 7. PMID 27388500
- [Background] Mduma E, Ersdal H, Svensen E, Kidanto H, Auestad B, Perlman J. Frequent brief on-site simulation training and reduction in 24-h neonatal mortality--an educational intervention study. Resuscitation. 2015 Aug;93:1-7. doi: 10.1016/j.resuscitation.2015.04.019. Epub 2015 May 6. PMID 25957942
- [Background] Arabi AM, Ibrahim SA, Ahmed SE, MacGinnea F, Hawkes G, Dempsey E, Ryan CA. Skills retention in Sudanese village midwives 1 year following Helping Babies Breathe training. Arch Dis Child. 2016 May;101(5):439-42. doi: 10.1136/archdischild-2015-309190. Epub 2016 Jan 29. PMID 26826172
- [Background] Wyckoff MH, Aziz K, Escobedo MB, Kapadia VS, Kattwinkel J, Perlman JM, Simon WM, Weiner GM, Zaichkin JG. Part 13: Neonatal Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S543-60. doi: 10.1161/CIR.0000000000000267. No abstract available. PMID 26473001
- [Background] FDIs, I. (2009). 9241-210 (2009). Ergonomics of human system interaction-Part 210: Human-centered design for interactive systems (formerly known as 13407). International Organization for Standardization (ISO). Switzerland.
- [Background] Krueger RA, Casey MA. Focus Groups: A practical guide for applied research. 4th ed. California: Sage Publications Inc., 2008.
- [Derived] Chan NH, Merali HS, Mistry N, Kealey R, Campbell DM, Morris SK, Data S. Development of a novel mobile application, HBB Prompt, with human factors and user-centred design for Helping Babies Breathe skills retention in Uganda. BMC Med Inform Decis Mak. 2021 Feb 4;21(1):39. doi: 10.1186/s12911-021-01406-z. PMID 33541340
- [Derived] Merali HS, Chan NH, Mistry N, Kealey R, Campbell D, Morris SK, Data S. Designing and evaluating a novel mobile application for Helping Babies Breathe skills retention in Uganda: comparative study protocol. BMJ Paediatr Open. 2019 Sep 3;3(1):e000561. doi: 10.1136/bmjpo-2019-000561. eCollection 2019. PMID 31549001

DOCUMENTS (1):
  • Study Protocol (2018-02-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT03577054/Prot_000.pdf